CLINICAL TRIAL: NCT00976989
Title: A Randomised, Multicentre, Multinational Phase II Study to Evaluate Pertuzumab in Combination With Trastuzumab, Given Either Concomitantly or Sequentially With Standard Anthracycline-based Chemotherapy or Concomitantly With a Non-anthracycline-based Chemotherapy Regimen, as Neoadjuvant Therapy for Patients With Locally Advanced, Inflammatory or Early Stage HER2-positive Breast Cancer
Brief Title: A Study of Pertuzumab in Combination With Herceptin and Chemotherapy in Participants With HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO22280; 2009-012019-17 (EudraCT Number)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Docetaxel

ARMS (3):
- T+P Concomitant Anthracycline-based chemotherapy (Experimental): 5-Fluorouracil, epirubicin with cyclophosphamide (FEC), trastuzumab (T) and pertuzumab (P) every three weeks for three cycles, followed by docetaxel, trastuzumab and pertuzumab every three weeks, for three cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 17 as adjuvant therapy post-surgery.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: FEC; Drug: Docetaxel
- T+P Sequential Anthracycline-based chemotherapy (Experimental): FEC every three weeks for three cycles, followed by docetaxel, trastuzumab (T) and pertuzumab (P) every three weeks, for three cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 21 as adjuvant therapy post-surgery.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: FEC; Drug: Docetaxel
- T+P Concomitant Non-Anthracycline chemotherapy (Experimental): Trastuzumab, carboplatin, docetaxel (TCH) and pertuzumab (P) every three weeks, for six cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 17 as adjuvant therapy post-surgery.
  Interventions: Drug: Pertuzumab; Drug: TCH

INTERVENTIONS:
Drug: Pertuzumab — 840 mg loading dose intravenously (IV), then 420 mg IV 3-weekly.
  Other Names: Perjeta
Drug: Trastuzumab — 8 mg/kg loading dose IV, then 6 mg/kg every 3 weeks.
  Other Names: Herceptin
  Arms: T+P Concomitant Anthracycline-based chemotherapy; T+P Sequential Anthracycline-based chemotherapy
Drug: FEC — 5-fluorouracil 500 mg/m^2, epirubicin 100 mg/m^2 and cyclophosphamide 600 mg/m^2.
  Arms: T+P Concomitant Anthracycline-based chemotherapy; T+P Sequential Anthracycline-based chemotherapy
Drug: Docetaxel — 75 mg/m^2 for the first dose; 100 mg/m^2 if no dose limiting toxicity occurs.
  Arms: T+P Concomitant Anthracycline-based chemotherapy; T+P Sequential Anthracycline-based chemotherapy
Drug: TCH — Trastuzumab followed by carboplatin at target area under the plasma concentration-time curve (AUC) 6 and docetaxel at a starting dose of 75 mg/m^2. All treatments were given every three weeks by the IV route.
  Arms: T+P Concomitant Non-Anthracycline chemotherapy

SUMMARY:
This 3 arm study will assess the tolerability, safety and efficacy of 3 neoadjuvant treatment regimens in participants with locally advanced, inflammatory or early stage human epidermal growth factor receptor 2 (HER2)-positive breast cancer. Before surgery, participants will be randomized to receive either A) 6 cycles of pertuzumab plus trastuzumab (Herceptin), with 5-fluorouracil/epirubicin/cyclophosphamide (FEC) for cycles 1-3 and docetaxel for cycles 4-6, or B) FEC for cycles 1-3 followed by pertuzumab plus trastuzumab with docetaxel for cycles 4-6, or C) 6 cycles of pertuzumab plus trastuzumab with docetaxel and carboplatin. Pertuzumab will be administered at a loading dose of 840 mg intravenously (iv), then 420 mg iv 3-weekly, trastuzumab at a loading dose of 8 mg/kg iv, then 6 mg/kg iv 3-weekly, docetaxel at 75 mg/m^2 iv, increased to 100 mg/m^2 iv 3-weekly, and FEC and carboplatin iv 3-weekly at standard doses. Following surgery participants will receive trastuzumab 6 mg/kg iv 3-weekly for a total of 1 year, as well as adequate chemo-, radio- and hormone therapy. Anticipated time on study treatment is 4-12 months, and target sample size is 200-300.

ELIGIBILITY:
Inclusion Criteria:

* female participants, age >/=18 years
* advanced, inflammatory or early stage unilateral invasive breast cancer
* HER2-positive breast cancer
* baseline left ventricular ejection fraction (LVEF) >/=55%

Exclusion Criteria:

* metastatic disease (Stage IV) or bilateral breast cancer
* previous anticancer therapy or radiotherapy for any malignancy
* other malignancy, except for carcinoma in situ of the cervix, or basal cell carcinoma
* clinically relevant cardiovascular disease
* current chronic treatment with corticosteroids of >10mg methylprednisolone or equivalent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo
- Brazil (2):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (3):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
- Pula, Croatia
- Germany (6):
  - Heidelberg
  - Kiel
  - Regensburg
  - Trier
  - Troisdorf
  - Ulm
- Greece (2):
  - Heraklion
  - Thessaloniki
- Italy (3):
  - Rome, Lazio
  - Monza, Lombardy
  - S. Fermo Della Battaglia (CO), Lombardy
- Mexico (2):
  - Mexico City
  - Xalapa
- Auckland, New Zealand
- Portugal (2):
  - Aveiro
  - Lisbon
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Belgrade, Serbia
- South Africa (2):
  - Durban
  - Pretoria
- South Korea (2):
  - Daegu
  - Seoul
- Spain (4):
  - Barcelona, Barcelona
  - Córdoba, Cordoba
  - Donostia / San Sebastian, Guipuzcoa
  - Madrid, Madrid
- Sweden (4):
  - Eskilstuna
  - Stockholm
  - Sundsvall
  - Umeå
- Switzerland (2):
  - Baden
  - Zurich
- Taiwan (2):
  - Taichung
  - Taipei
- Nassau, The Bahamas
- United Kingdom (7):
  - Bournemouth
  - Derby
  - Guildford
  - Newcastle upon Tyne
  - Southampton
  - Truro
  - Westcliffe-on-sea

REFERENCES:
- [Derived] Schneeweiss A, Chia S, Hickish T, Harvey V, Eniu A, Waldron-Lynch M, Eng-Wong J, Kirk S, Cortes J. Long-term efficacy analysis of the randomised, phase II TRYPHAENA cardiac safety study: Evaluating pertuzumab and trastuzumab plus standard neoadjuvant anthracycline-containing and anthracycline-free chemotherapy regimens in patients with HER2-positive early breast cancer. Eur J Cancer. 2018 Jan;89:27-35. doi: 10.1016/j.ejca.2017.10.021. Epub 2017 Dec 8. PMID 29223479
- [Derived] Swain SM, Schneeweiss A, Gianni L, Gao JJ, Stein A, Waldron-Lynch M, Heeson S, Beattie MS, Yoo B, Cortes J, Baselga J. Incidence and management of diarrhea in patients with HER2-positive breast cancer treated with pertuzumab. Ann Oncol. 2017 Apr 1;28(4):761-768. doi: 10.1093/annonc/mdw695. PMID 28057664
- [Derived] Schneeweiss A, Chia S, Hegg R, Tausch C, Deb R, Ratnayake J, McNally V, Ross G, Kiermaier A, Cortes J. Evaluating the predictive value of biomarkers for efficacy outcomes in response to pertuzumab- and trastuzumab-based therapy: an exploratory analysis of the TRYPHAENA study. Breast Cancer Res. 2014 Jul 8;16(4):R73. doi: 10.1186/bcr3690. PMID 25005255
- [Derived] Schneeweiss A, Chia S, Hickish T, Harvey V, Eniu A, Hegg R, Tausch C, Seo JH, Tsai YF, Ratnayake J, McNally V, Ross G, Cortes J. Pertuzumab plus trastuzumab in combination with standard neoadjuvant anthracycline-containing and anthracycline-free chemotherapy regimens in patients with HER2-positive early breast cancer: a randomized phase II cardiac safety study (TRYPHAENA). Ann Oncol. 2013 Sep;24(9):2278-84. doi: 10.1093/annonc/mdt182. Epub 2013 May 22. PMID 23704196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 3 periods: Neoadjuvant (pre-operative) period and surgery, adjuvant (post-operative) period and post-treatment follow-up period.
Groups:
- T+P Concomitant Anthracycline-based Chemotherapy: 5-Fluorouracil, epirubicin with cyclophosphamide (FEC), trastuzumab and pertuzumab every three weeks for three cycles, followed by docetaxel, trastuzumab and pertuzumab every three weeks, for three cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 17 as adjuvant therapy post-surgery.
- T+P Sequential Anthracycline-based Chemotherapy: FEC every three weeks for three cycles, followed by docetaxel, trastuzumab and pertuzumab every three weeks, for three cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 21 as adjuvant therapy post-surgery.
- T+P Concomitant Non-Anthracycline Chemotherapy: Trastuzumab, carboplatin, docetaxel (TCH) and pertuzumab every three weeks, for six cycles as neoadjuvant therapy. Trastuzumab every three weeks from Cycle 7 up to Cycle 17 as adjuvant therapy post-surgery.
Period: Overall Study
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Started | 73 | 75 | 77
Completed | 60 | 63 | 60
Not Completed | 13 | 12 | 17
Not completed — Violation of Selection Criteria at Entry | 1 | 0 | 1
Not completed — Death | 5 | 7 | 10
Not completed — Refused Treatment | 4 | 3 | 5
Not completed — Failure to Return | 2 | 1 | 0
Not completed — Recurrence of Disease | 0 | 1 | 0
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy | Total
Number analyzed (Participants) | 73 | 75 | 77 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.41) | 50.5 (10.70) | 50.6 (10.58) | 50.6 (10.86)
Gender [Count of Participants; unit: Participants]
  Female | 73 | 75 | 77 | 225
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety: Percentage of Participants With Symptomatic Cardiac Events as Assessed by the Investigator
Description: Left ventricular systolic dysfunction (LVSD) as assessed by the Investigator, including Grade 3, 4 or 5 symptomatic LVSD with symptomatic cardiac events.
Time Frame: From baseline up to approximately 3.5 years
Population: Safety population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 72 | 75 | 76
percentage of participants | 0 | 2.7 | 1.3

2. Primary Outcome: Safety: Percentage of Participants With Left Ventricular Ejection Fraction (LVEF) Decline During Pre-operative (Neoadjuvant) Period
Description: Percentage of participants with LVEF measures decline of ≥ 10% from baseline and to a value of <50% during the pre-operative (neoadjuvant) period.
Time Frame: From baseline up to approximately 18 weeks
Population: Safety population included all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 72 | 75 | 76
percentage of participants | 5.6 | 5.3 | 3.9

3. Secondary Outcome: Efficacy: Percentage of Participants With Complete Pathological Response (pCR)
Description: pCR is defined as the absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy. pCR is evaluated after 6 cycles of treatment and surgery or following withdrawal from the study whichever occurs sooner.
Time Frame: At surgery, after 18 weeks (6 cycles) of treatment
Population: Intent to treat (ITT) population included all participants who were randomized to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 73 | 75 | 77
percentage of participants | 61.6 [49.5 to 72.8] | 57.3 [45.4 to 68.7] | 66.2 [54.6 to 76.6]

4. Secondary Outcome: Efficacy: Clinical Response Rate
Description: Tumor response is defined as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) and is identified as per local practice. Clinical response rate is defined as the percentage of participants who achieve a response of CR or PR at any time pre-surgery. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by mammogram or magnetic resonance imaging (MRI) and clinical breast examination (CBE), CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: During each 3-week cycle of 6 total cycles: up to 18 weeks
Population: ITT population included all participants who were randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 73 | 75 | 77
percentage of participants | 91.8 | 94.7 | 89.6

5. Secondary Outcome: Efficacy: Time to Clinical Response
Description: Time to clinical response is defined as the time from the date of first dose received to the first date of assessment of clinical response. Clinical response is defined as a response of CR or PR at any time pre-surgery. Per RECIST v1.0 for target lesions and assessed by mammogram or MRI and CBE, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 18 weeks
Population: ITT population included all participants who were randomized to treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 73 | 75 | 77
weeks | 3.6 [3 to 6] | 6.3 [6 to 7] | 4.9 [4 to 6]

6. Secondary Outcome: Efficacy: Percentage of Participants Achieving Breast Conserving Surgery
Description: This is the percentage of participants who achieved breast conserving surgery out of the intent-to-treat population without inflammatory breast cancer, as these participants received mastectomy irrespective of their response to neoadjuvant (pre-operative) treatment.
Time Frame: At approximately 18 weeks
Population: Number of participants analyzed represents the participants with T2-3 tumors for whom mastectomy was planned.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 46 | 36 | 37
percentage of participants | 21.7 | 16.7 | 27.0

7. Secondary Outcome: Efficacy: Percentage of Participants Without an Overall Survival (OS) Event
Description: Overall survival (OS) was defined as the time from randomization to the date of death from any cause. Participants who were alive or lost to follow-up were censored at the last known alive date. Participants with no post-baseline information were censored at the date of randomization plus one day.
Time Frame: From baseline to end of study up to 5 years
Population: ITT population included all participants who were randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 73 | 75 | 77
percentage of participants | 93.2 | 90.7 | 87.0

8. Secondary Outcome: Efficacy: Percentage of Participants Without a Disease-Free Survival (DFS) Event
Description: The DFS was defined as the time from the first date of no disease (i.e., date of surgery) to the first documentation of progressive disease (PD) or death. PD was assessed using RECIST v1.0 and MRI and CBE. It was defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions. Any evidence of contralateral disease in situ was not considered as PD. Participants who were withdrawn from the study without documented PD were censored at the date of the last assessment when the participant was known to be disease-free.
Time Frame: From baseline to end of study up to 5 years
Population: ITT population included all participants who were randomized to treatment. Number of participants analyzed is total number of participants evaluable during each period.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 69 | 67 | 72
percentage of participants | 85.5 | 88.1 | 84.7

9. Secondary Outcome: Efficacy: Percentage of Participants Without a Progression-Free Survival (PFS) Event
Description: Progression-free survival was defined as the time from the date of randomization to the first documentation of PD or death from any cause, whichever occurred first. PD was assessed using RECIST v1.0 and MRI and CBE. It was defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions. Participants who were withdrawn from the study without documented PD were censored at the date of the last assessment when the participant was known to be free from PD. Participants without post-baseline assessments but known to be alive were censored at the time of randomization plus one day.
Time Frame: From baseline to end of study up to 5 years
Population: ITT population included all participants who were randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 73 | 75 | 77
percentage of participants | 86.3 | 85.3 | 81.8

10. Secondary Outcome: Safety: Percentage of Participants With Cardiac Symptoms Associated With Symptomatic Left Ventricular Systolic Dysfunction (LVSD)
Description: Percentage of participants with signs or symptoms of cardiac events.
Time Frame: From Baseline to end of Neoadjuvant Period (up to 18 weeks), Adjuvant Period (up to 1.5 years), Follow-up Period (up to 3.5 years)
Population: Safety analysis population included all randomized participants who received treatment. Number of participants analyzed is total number of participants evaluable during each period.
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 72 | 75 | 76
percentage of participants
  Neoadjuvant Period (n=72, 75, 76) | 1.4 | 2.7 | 0
  Adjuvant Period (n= 68, 65, 67) | 0 | 0 | 1.5
  Follow-up Period (n=70, 75, 74) | 0 | 1.3 | 0

11. Secondary Outcome: Safety: Percentage of Participants With Asymptomatic Left Ventricular Ejection Fraction (LVEF) Events
Description: Percentage of participants with LVEF events without signs or symptoms of cardiac events.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 72 | 75 | 76
percentage of participants
  Neoadjuvant Period (n=72, 75, 76) | 5.6 | 4.0 | 2.6
  Adjuvant Period (n= 66, 64, 63) | 3.0 | 0 | 4.8
  Follow-up Period (n=21, 18, 23) | 0 | 11.1 | 4.3

12. Secondary Outcome: Safety: Maximum Decrease in Left Ventricular Ejection Fraction (LVEF) Measures
Description: Maximum decrease in LVEF measures is the change from baseline at worst treatment value. LVEF is measured as percentage.
Time Frame: From baseline up to approximately 3.5 years
Population: Safety analysis population included all randomized participants who received treatment. Number of participants analyzed is total number of participants evaluable.
Measure: Mean (Standard Deviation); unit: percentage (ejection fraction)
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Number analyzed (Participants) | 71 | 72 | 73
percentage (ejection fraction) | -6.6 (5.15) | -8.4 (5.66) | -7.0 (6.48)

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: Safety population included all participants who were randomized and received study drug.
Arm/Group | T+P Concomitant Anthracycline-based Chemotherapy | T+P Sequential Anthracycline-based Chemotherapy | T+P Concomitant Non-Anthracycline Chemotherapy
Serious Adverse Events (participants affected / at risk) | 23/72 | 18/75 | 31/76
Other Adverse Events (participants affected / at risk) | 72/72 | 73/75 | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T+P Concomitant Anthracycline-based Chemotherapy (N=72) | T+P Sequential Anthracycline-based Chemotherapy (N=75) | T+P Concomitant Non-Anthracycline Chemotherapy (N=76)
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 | 4 | 11
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 2
Neutropenic infection (Infections and infestations) | 0 | 2 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Lung Abscess (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 3 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Breast necrosis (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T+P Concomitant Anthracycline-based Chemotherapy (N=72) | T+P Sequential Anthracycline-based Chemotherapy (N=75) | T+P Concomitant Non-Anthracycline Chemotherapy (N=76)
Diarrhoea (Gastrointestinal disorders) | 46 | 44 | 55
Nausea (Gastrointestinal disorders) | 38 | 41 | 34
Vomiting (Gastrointestinal disorders) | 29 | 27 | 30
Dyspepsia (Gastrointestinal disorders) | 19 | 9 | 17
Constipation (Gastrointestinal disorders) | 14 | 18 | 13
Stomatitis (Gastrointestinal disorders) | 10 | 13 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 6
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 8
Haemorrhoids (Gastrointestinal disorders) | 5 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 4
Oral pain (Gastrointestinal disorders) | 1 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 39 | 42
Rash (Skin and subcutaneous tissue disorders) | 17 | 8 | 20
Nail disorder (Skin and subcutaneous tissue disorders) | 9 | 8 | 10
Erythema (Skin and subcutaneous tissue disorders) | 10 | 5 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 7 | 8
Palmar -plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 9 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7 | 4
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 5 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Fatigue (General disorders) | 30 | 28 | 33
Mucosal inflammation (General disorders) | 17 | 15 | 12
Pyrexia (General disorders) | 11 | 9 | 15
Asthenia (General disorders) | 9 | 14 | 10
Oedema peripheral (General disorders) | 10 | 5 | 9
Pain (General disorders) | 3 | 7 | 4
Chills (General disorders) | 4 | 1 | 7
Chest pain (General disorders) | 2 | 4 | 5
Influenza like illness (General disorders) | 2 | 5 | 2
Oedema (General disorders) | 1 | 3 | 5
Malaise (General disorders) | 0 | 2 | 5
Axillary pain (General disorders) | 0 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 36 | 33 | 37
Anaemia (Blood and lymphatic system disorders) | 14 | 8 | 29
Leukopenia (Blood and lymphatic system disorders) | 16 | 12 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 18 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 16 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2
Headache (Nervous system disorders) | 20 | 15 | 16
Dysgeusia (Nervous system disorders) | 8 | 10 | 16
Dizziness (Nervous system disorders) | 7 | 9 | 15
Neuropathy peripheral (Nervous system disorders) | 5 | 4 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 8 | 5
Paraesthesia (Nervous system disorders) | 3 | 4 | 9
Polyneuropathy (Nervous system disorders) | 4 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7
Nasopharyngitis (Infections and infestations) | 6 | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 7 | 10 | 3
Urinary tract infection (Infections and infestations) | 5 | 7 | 7
Rhinitis (Infections and infestations) | 6 | 1 | 4
Cystitis (Infections and infestations) | 0 | 4 | 6
Insomnia (Psychiatric disorders) | 12 | 13 | 17
Depression (Psychiatric disorders) | 3 | 3 | 4
Anxiety (Psychiatric disorders) | 1 | 4 | 4
Hot Flush (Vascular disorders) | 11 | 9 | 10
Hypertension (Vascular disorders) | 5 | 2 | 5
Lymphoedema (Vascular disorders) | 2 | 5 | 4
Haemoglobin decreased (Investigations) | 6 | 4 | 7
Alanine aminotransferase increased (Investigations) | 5 | 3 | 8
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 5
Weight decreased (Investigations) | 3 | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 15 | 8 | 16
Radiation skin injury (Injury, poisoning and procedural complications) | 11 | 14 | 7
Seroma (Injury, poisoning and procedural complications) | 4 | 4 | 1
Lacrimation increased (Eye disorders) | 9 | 4 | 6
Conjunctivitis (Infections and infestations) | 3 | 2 | 4
Eyelid oedema (Eye disorders) | 1 | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 7 | 8 | 7
Palpitations (Cardiac disorders) | 3 | 1 | 4
Breast pain (Reproductive system and breast disorders) | 2 | 3 | 6
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 4
Drug hypersensitivity (Immune system disorders) | 6 | 2 | 7
Dysuria (Renal and urinary disorders) | 2 | 0 | 7
Influenza (Infections and infestations) | 5 | 4 | 2
Chest discomfort (General disorders) | 4 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.